CLINICAL TRIAL: NCT04995653
Title: A Phase 1b Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of SER-155 in Adults Undergoing Hematopoietic Stem Cell Transplantation (HSCT) to Reduce the Risk of Infection and Graft vs. Host Disease (GvHD)
Brief Title: A Multiple Dose Study to Evaluate Safety, Tolerability, PK, and Efficacy of SER-155 in Adults Undergoing HSCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seres Therapeutics, Inc. (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SER-155-001
Record Dates: First submitted 2021-07-13; First posted 2021-08-09 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation
Keywords: Microbiome; stem cell transplant

STUDY DESIGN:
Intervention Model Description: There are 2 parts or cohorts for the trial. Cohort 1 is an open-label study. Cohort 2 is double-blind, randomized, placebo-controlled study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Open Label Study (Experimental): Vancomycin & SER-155
  Interventions: Drug: Vancomycin Pre-Treatment; Drug: SER-155
- Cohort 2 - Randomized, Double-Blind, Placebo-Controlled Study (Experimental): Vancomycin & SER-155 OR Vancomycin placebo & SER-155 placebo
  Interventions: Drug: Vancomycin Pre-Treatment; Drug: Vancomycin Placebo; Drug: SER-155; Drug: SER-155 Placebo

INTERVENTIONS:
Drug: Vancomycin Pre-Treatment — Four times daily dosing with Vancomycin
Drug: Vancomycin Placebo — Four times daily dosing with Vancomycin Placebo
  Arms: Cohort 2 - Randomized, Double-Blind, Placebo-Controlled Study
Drug: SER-155 — Once daily dosing with SER-155
Drug: SER-155 Placebo — Once daily dosing with SER-155 placebo
  Arms: Cohort 2 - Randomized, Double-Blind, Placebo-Controlled Study

SUMMARY:
An Open-Label and Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of SER-155 in Adults Undergoing Hematopoietic Stem Cell Transplantation to Reduce the Risk of Infection and Graft vs. Host Disease

DETAILED DESCRIPTION:
This is a Phase 1b randomized, double-blind, placebo-controlled, multiple dose, multicenter study designed to evaluate the safety, efficacy, and microbiome alterations associated with SER-155 dosing, after microbiome conditioning with oral vancomycin, in adult subjects aged ≥18 years who are undergoing Hematopoietic Stem Cell Transplantation (HSCT).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥ 18 years of age undergoing HSCT.
* Planning to undergo allogeneic hematopoietic stem cell transplantation from a human leukocyte antigen matched related donor, haploidentical related donor, HLA-matched unrelated donor, or HLA 1-antigen mismatched unrelated or related donor, with either bone marrow or peripheral blood stem cells as a graft source, and with any conditioning regimen

Exclusion Criteria:

* Severe colitis of any etiology or active/currently-treated inflammatory bowel disease (IBD) or total colectomy.
* Evidence of relapse or progression of hematologic malignancy (minimal residual disease is allowed).
* Transplant using umbilical cord blood or ex vivo T-cell-depleted HSCT
* Receipt of chimeric antigen receptor T-cell (CAR-T) therapy.
* Received a fecal microbiota transplant (FMT) or any live microbial therapeutic within 3 months prior to Screening.
* Known allergy or intolerance to oral vancomycin.
* Concomitant participation or participation within 14 days or 5 half-lives of another investigational unapproved treatment, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SER-155, including incidence and severity of adverse events, serious adverse events, or adverse events of special interest | Day 100
  Incidence and severity of participants with adverse events, serious adverse events, or adverse events of special interest
Engraftment of SER-155 | Day 100
  Prevalence of SER-155 strains in subject stool measured before and after treatment courses

SECONDARY OUTCOMES:
Abundance of Enterococcus and Enterobacteriaceae | Day 100
Combined and individual incidence of bloodstream infections, gastrointestinal infections, and acute Graft-versus Host Disease | Day 100
Incidence and duration of febrile neutropenia | Day 100

CONTACTS AND LOCATIONS:
Overall Officials: Doris Ponce, MD, Principal Investigator — MSKCC; Bina Tejura, MD, Study Director — Seres Therapeutics, Inc.
Locations (13):
- United States (13):
  - Banner Health - MD Anderson Medical Center, Gilbert, Arizona
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - University of California, Los Angeles - Division of Hematology-Oncology, Marina del Rey, California
  - Georgetown (MedStar Health), Washington D.C., District of Columbia
  - University of Florida - Division of Hematology & Oncology, Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Harvard Medical School - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No